CLINICAL TRIAL: NCT03863171
Title: Early Diagnosis for Ocular Ischemia Syndrome Using Arterial Spin Labeling Magnetic Resonance Imaging Technique: a Prospective Multicenter Cohort Study
Brief Title: Early Diagnosis for Ocular Ischemia Syndrome Using Arterial Spin Labeling Magnetic Resonance Imaging Technique
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Yue Li, Clinical Professor, Beijing Friendship Hospital
Other Study IDs: 2018-P2-185-02
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Ocular Ischemia Syndrome
MeSH Terms: interventions — Magnetic Resonance Imaging; Fluorescein Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ocular ischemia syndrome: Patients with ocular ischemia syndrome
  Interventions: Diagnostic Test: Arterial spin labeling (ASL) magnetic resonance imaging; Diagnostic Test: Fundus fluorescein angiography
- Control: Patients with age-related macular degeneration
  Interventions: Diagnostic Test: Arterial spin labeling (ASL) magnetic resonance imaging; Diagnostic Test: Fundus fluorescein angiography

INTERVENTIONS:
Diagnostic Test: Arterial spin labeling (ASL) magnetic resonance imaging — Arterial spin labeling (ASL) magnetic resonance imaging test
Diagnostic Test: Fundus fluorescein angiography — Fundus fluorescein angiography test

SUMMARY:
1. To evaluate ocular blood perfusion status and the possibility of craniocerebral vascular lesions of patients with ocular ischemia syndrome (OIS) using arterial spin labeling (ASL) magnetic resonance imaging technique.
2. To evaluate the specificity, sensitivity and accuracy of arterial spin labeling (ASL) magnetic resonance imaging technique in OIS diagnosis, compared with the traditional routine examination method.

ELIGIBILITY:
Inclusion Criteria:

* Ocular ischemia syndrome group: Patients diagnosed with ocular ischemia syndrome;
* Age-related macular degeneration group (Control group): Patients diagnosed with age-related macular degeneration;
* Age: 50-80 years;
* Sex: all;
* Patients signed written informed consent.

Exclusion Criteria:

* Fundus fluorescein angiography (FFA) clear images cannot be obtained due to refractive media problems(such as corneal leukoplakia, severe cataract, vitreous hemorrhage, etc.) ;
* Patients with contraindications for FFA;
* Patients was unable to perform magnetic resonance rmaging (MRI) test;
* Patients with history of bleeding and cerebral infarction;
* Patients with a history of surgery within 3 months;
* Patients who had participated in other clinical trials within 3 months;
* Patients who disagree and refuse to participate in the trial.

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with ocular ischemia syndrome
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Blood Flow (BF) | through study completion, an average of 2 years
  Blood Flow (BF)：a parameter measured by arterial spin labeling perfusion MRI to qualify the perfusion in tissue-specific units (ml blood/gram tissue/time)

CONTACTS AND LOCATIONS:
Overall Officials: Yanling Wang, MD, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China